CLINICAL TRIAL: NCT06480825
Title: Ulta-High Frequency Ultrasound Assessment of Normal Versus Gingivitis Affected Gingival Tissues
Brief Title: Application of Ultra-high Frequency Ultrasonography (UHFUS) to the Study of Gingival Tissues
Status: Recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Rossana Izzetti, Principal Investigator, Researcher at the Department of Surgical, Medical and Molecular Pathology and Critical Care Medicine of the University of Pisa, University of Pisa
Other Study IDs: 7935870439
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Gingivitis; Periodontitis
MeSH Terms: conditions — Gingivitis; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gingivitis group: patients affected by gingivitis
  Interventions: Other: Performance of ultrasonographic scan
- Control group: Periodontally healthy patients
  Interventions: Other: Performance of ultrasonographic scan

INTERVENTIONS:
Other: Performance of ultrasonographic scan — Ultra-high frequency ultrasonographic scan of gingival tissues

SUMMARY:
Gingival inflammation triggered by the accumulation of bacterial is the primary risk factor for the development of periodontitis. Clinically, localized signs of inflammation limited to the gingiva, presence of significant bacterial plaque load, and stable attachment levels on the periodontium can be observed in course of gingivitis. The aim of the present study is to compare clinical aspects of gingival tissue in healthy patients versus patients with gingivitis to assess the ultrastructural variations present in course of inflammation.

Patients with gingivitis and healthy controls will be enrolled. All patients will undergo ultra-high frequency ultrasonographic scans (70 MHz) of gingival tissue on three areas per dental arch (anterior, middle right, middle left). Gingival thickness, echogenicity, and vascularization assessed through resisitive index will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* males or females of age > 18 years
* presence of at least 20 teeth
* full-mouth plaque score (FMPS) >50%
* FMBS >30%
* ability and willingness to give informed consent

Exclusion Criteria:

* pregnancy or breastfeeding
* pharmacological treatment with antinflammatory drugs, statins, or either local or systemic antibiotics (within the previous 30 days)
* smoking habit
* dental or periodontal condition requiring immediate treatment
* refusal to be enrolled in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to the Sub-Unit of Periodontology, Halitosis, and Periodontal Medicine of the Unit of Dentistry and Oral Surgery at the University Hospital of Pisa will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Echogenicity | measured once at enrollemnt
  Variations in echogenicity assessed through grey levels distribution between healthy patients versus gingivitis

SECONDARY OUTCOMES:
Vascular parameters | measured once at enrollemnt
  Variations in vascularization assessed through grey levels distribution between healthy patients versus gingivitis
DMFT | measured once at enrollement
  The Decayed-Missing-Filled Teeth (DMFT) index, categorized as Low (0-4), Moderate (5-13), and High (14+), will evaluate overall dental health.
PPD | measured once at enrollement
  Probing Pocket Depth (PPD) will be measured using a UNC-15 periodontal probe with 0.3 N pressure, recording six sites per tooth (distobuccal, buccal, mesiobuccal, distolingual, lingual, mesiolingual), rounded to the nearest millimeter.
FMBS | measured once at enrollement
  Full Mouth Bleeding Score (FMBS) will be determined dichotomously post-probing.
FMPS | measured once at enrollement
  Full Mouth Plaque Score (FMPS) will assess plaque presence on each tooth surface, with scores of 1 for presence and 0 for absence across six sites per tooth.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University of Pisa, Pisa
  - Department of Surgical, Medical and Molecular Pathology and Critical Care Medicine, University Hospital of Pisa, Pisa